CLINICAL TRIAL: NCT05025956
Title: The Use of Senolytic Agent to Improve the Benefit of Platelet-Rich Plasma and Losartan for Treatment of Femoroacetabular Impingement and Labral Tear: A Pilot Study
Brief Title: Senolytic Agent Improve the Benefit of Platelet-Rich Plasma and Losartan
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Steadman Philippon Research Institute (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-058
Record Dates: First submitted 2021-08-02; First posted 2021-08-30 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Femoroacetabular Impingement
Keywords: FAI Labral tear Fisetin Losartan
MeSH Terms: conditions — Femoracetabular Impingement | interventions — fisetin

STUDY DESIGN:
Intervention Model Description: pilot, prospective, randomized, double-blind, placebo control clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Investigator or properly trained and delegated study team member (research PA) will write the prescription for the study medication. The subject's randomization block and within-block random number will be communicated directly to the Vail Health pharmacy. The Vail Health pharmacy will maintain an unblinded, de-identified randomization spreadsheet that documents group allocation for each subject. The Vail Health Pharmacy oversees and manages drug disbursement for research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fisetin group (investigational group) (Experimental): 20mg/kg of Fisetin per day for days 1 and 2 prior to surgery and days 33, 34, 63, 64, 93, and 94 post surgery.
  (The pills are 100mg each. For example, if a participant weighs 160 pounds (about 73 kg), the participant will need to take 15 pills per day)
  Interventions: Drug: Fisetin
- Placebo group (control group) (Placebo Comparator): 20mg/kg of Placebo per day for days 1 and 2 prior to surgery and days 33, 34, 63, 64, 93, and 94 post surgery.
  (The pills are 100mg each. For example, if a participant weighs 160 pounds (about 73 kg), the participant will need to take 15 pills per day)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fisetin — Oral Fisetin 20 mg/kg taken for 8 days total.
  Other Names: Novusetin; 7,3',4'-flavon-3-ol; 3,3',4',7-tetrahydroxyflavone
  Arms: Fisetin group (investigational group)
Drug: Placebo — Fisetin appearance-matched microcrystalline cellulose placebo. 20 mg/kg taken for 8 days total.
  Other Names: Placebo Oral Capsule
  Arms: Placebo group (control group)

SUMMARY:
The purpose is to explore the possible benefit of administration of Fisetin, (a senolytic agent) to improve the benefit of Platelet-Rich Plasma and losartan for treatment of femoroacetabular impingement and labral tear.

We believe that giving Fisetin, a senolytic agent, will improve the benefit of PRP by eliminating senescent cells and senescence-associated secretory phenotype (SASP), known to exist in PRP. The main objectives of this study are to determine if pre- and post-operative administration of a senolytic agent will improve the beneficial effects of PRP when used in conjunction with surgical treatment of FAI and/or labral tear, to determine whether pre- and postoperative administration of Fisetin is associated with adverse events, and to determine if pre- and post-operative administration of Fisetin leads to a decrease in systemic senescence, serum SASP, and fibrotic markers.

Patients suffering from femoroacetabular impingement and labral tear, who are planning to undergo hip arthroscopy combined with standard of care intra-operative PRP injection and post-operative losartan administration will be recruited from the clinical practice of the Principal Clinical Investigator or his designee at The Steadman Clinic (TSC).

DETAILED DESCRIPTION:
This is a pilot, prospective, randomized, double-blind, placebo control clinical trial is proposed to evaluate the safety and efficacy of a senolytic agent (Fisetin) to improve the benefits of standard of care platelet rich plasma (PRP) injection and antifibrotic medication (Losartan) in patients undergoing hip arthroscopy for treatment of femoroacetabular impingement (FAI) and/or labral tear (LT).

ELIGIBILITY:
Inclusion Criteria:

* Capacity to personally give informed consent (consent via legally authorized representative will not be accepted) and who are willing to comply with all study-related procedures and assessments
* Between 18 and 80 years of age
* Have been diagnosed with femoroacetabular impingement (FAI) and/or a hip labral tear
* You are scheduled to undergo hip arthroscopy to treat FAI and /or a hip labral tear

Exclusion Criteria:

* Previous or Planned Hip Surgeries, Procedures and/or Treatments:
* Planned surgery on either the contralateral or target hip at any time during the Study period including dosing and follow-up
* Require microfracture on the target hip as part of the planned arthroscopy
* Within 6 months of signing informed consent, has undergone regenerative hip joint procedures on the target hip including, but not limited to, platelet-rich plasma injections, mesenchymal stem cell transplantation
* Have had previous surgery (including microfracture) or diagnostic arthroscopy on the target hip
* Joint space less than ≤2mm
* Tönnis Grade 2-3
* Have a history of pigmented villonodular synovitis (joint disease characterized by inflammation and overgrowth of the synovial lining of the hip joint)
* Have a history of synovial chondromatosis (noncancerous tumor that develops in the synovial lining of the hip joint);
* Have a history of hip dysplasia requiring PAO
* History of Avascular Necrosis (AVN), Perthes disease, or slipped capital femoral epiphysis (SCFE)
* Any active known or suspected systemic autoimmune disease (except for vitiligo, residual auto-immune hypothyroidism requiring hormone replacement only, psoriasis not requiring systemic treatment for two years, conditions not expected to recur in the absence of an external trigger) or any history of a systemic inflammatory arthritis such as psoriatic, rheumatoid, ankylosing spondylitis or reactive arthritis
* Current diagnosis of fibromyalgia based on ACR criteria
* Are unable to or are unwilling to receive a PRP injection as part of your surgery
* Inadequate amount of PRP collected to serve the needs of the patient, and/or ProofPoint Biologics
* Within 2 years of signing informed consent, history of active blood clotting disorders requiring preventative treatment, or active malignancy of any type or history of a malignancy (with the exception of subjects with a history of treated basal or squamous cell carcinoma)
* Baseline HbA1C greater than 6.5, uncontrolled diabetes mellitus, and/or medication management has not been stable in the previous 2 months
* Current or prior history of other joint diseases that may (in the opinion of the Principal Clinical Investigator or his/her designee) confound study data or increase Subject risk. These may include including but not limited to joint dysplasia, crystal-induced arthropathy (such as gout, or calcium pyrophosphate deposition disease evidenced by clinical and/or radiographic means), aseptic osteonecrosis, acromegaly, Paget's disease, Ehlers-Danlos Syndrome, Gaucher's disease, Stickler syndrome, joint infection, hemochromatosis, or neuropathic arthropathy of any cause
* Any medical condition, including findings in laboratory or medical history or in the baseline assessments, that (in the opinion of the Principal Clinical Investigator or his/her designee), constitutes a risk or contraindication for participation in the Study or that could interfere with the Study conduct, endpoint evaluation or prevent the subject from fully participating in all aspects of the Study
* Females who are nursing a child, are pregnant, or who are planning to become pregnant during study drug dosing, or who are not willing to abstain from sex without the use of contraceptive protection during study drug dosing
* Males who do not wish to abstain from sex with women of childbearing potential without use of contraceptive protection during study drug dosing
* Currently taking warfarin or any drug that could cause a coagulopathy event
* Within 1 week of signing informed consent. taking medications that affect insulin activity, including Metformin or Acarbose
* Have an allergy to any active or inactive ingredient of Losartan or Fisetin, and/or currently taking medication with known adverse Losartan or Fisetin interaction
* Within 3 months of signing informed consent have taken senolytic agents including: Fisetin, Quercetin, Luteolin, Dasatinib, Piperlongumine, or Navitoclax;
* Currently taking the following drugs if they cannot be held for at least 2 days (per enrolling Principal Investigator or Sub Investigator, or healthcare professional appropriately delegated by the Principal Investigator) before and during administration of Fisetin: cyclosporine, tacrolimus, repaglinide, and bosentan
* Currently taking drugs that induce cellular senescence, including alkylating agents, anthracyclines, platins, other chemotherapy
* Within 1 month of signing informed consent, taking a glucocorticoid
* Has current history of drug and/or alcohol abuse
* Within the 3 months of signing informed consent has received anticonvulsant therapy, pharmacological doses of thyroid hormone (causing decline of thyroid stimulating hormone below normal)
* Within the 12 months prior to signing informed consent received any medications that affect bone turnover, including: adrenocorticosteroids (> 3 months at any time or > 10 days, estrogen (E) therapy or treatment with a selective E receptor modulator, or teriparatide
* Inability to tolerate oral medication.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-10-24 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | From date of study drug dosing until the end of the study, an average of 12 months
  Occurrence of adverse events

SECONDARY OUTCOMES:
Patient Reported Outcomes Questionnaire-Modified Harris Hip Score (mHHS) | Baseline, 8-12 weeks post-op, 6 months post-op, and 12 months post-op
  Consists of 8 questions covering domains of pain, gait, and functional activities. Scored on a 100-point scale, with each answer receiving a specific amount of points. Higher score represents greater hip health.
Patient Reported Outcomes Questionnaire- Hip Outcome Score: activities of daily living and sports subscales (HOS-ADL, HOS-SSS) | Baseline, 8-12 weeks post-op, 6 months post-op, and 12 months post-op
  Includes two subscales to calculate the total score:19 items in the HOS-ADL subscale and 9 items in the HOS-sports subscale.
Patient Reported Outcomes Questionnaire-Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Baseline, 8-12 weeks post-op, 6 months post-op, and 12 months post-op
  Scale from 0-96. Higher score represents worse hip health.
Patient Reported Outcomes Questionnaire-Optum Short Form physical and mental component scores (SF-12 PCS and SF-12 MCS) | Baseline, 8-12 weeks post-op, 6 months post-op, and 12 months post-op
  Includes two subscales to calculate the total score. Higher score represents greater health. Scale standardized to a US Population mean of 50 and standard deviation of 10 points.
Patient Reported Outcomes Questionnaire-Tegner Activity Scale | Baseline, 8-12 weeks post-op, 6 months post-op, and 12 months post-op
  Scale from 0-10. Higher score represents greater activity level.
Patient Reported Outcomes Questionnaire-Numeric Rating Scale for Hip Pain | Baseline, 8-12 weeks post-op, 6 months post-op, and 12 months post-op
  Scale from 1-10. Higher score represents greater hip pain.
Patient Reported Outcomes Questionnaire-Patient satisfaction with surgical outcome | Baseline, 8-12 weeks post-op, 6 months post-op, and 12 months post-op
  1-10-point scale
Multi and singleplex immunoassays and flow cytometry senescence and SASP marker assessment of peripheral blood | Baseline, and 8-12 weeks post-op
  Concentrations of secreted protein markers found in serum in pg/ml
Incidence of revision arthroscopy or other hip surgery required post initial arthroscopy | From day of initial surgery until the end of the study, an average of 12 months
  Incidence of revision surgery from day of initial surgery will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Johnny L Huard, PhD, Principal Investigator — Steadman Philippon Research Institute
Locations (1):
- The Steadman Clinic, Vail, Colorado, United States

IPD SHARING:
Plan to Share IPD: No